CLINICAL TRIAL: NCT04621565
Title: Withholding Hydrocortisone vs Routine Use of Hydrocortisone During Peri-operation in Pituitary Adenoma Patients With Intact Hypothalamus-Pituitary-Adrenal Axis: Randomized Controlled Trial to Assess Safety and Complications
Brief Title: Hydrocortisone Use During Peri-operation for Pituitary Adenomas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ZS-2608
Record Dates: First submitted 2020-10-28; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Pituitary Adenoma; Adrenal Insufficiency; Surgery
Keywords: Pituitary Adenomas; Peri-operation; Hydrocortisone; Adrenal Insufficiency
MeSH Terms: conditions — Pituitary Neoplasms; Adrenal Insufficiency | interventions — Saline Solution; Hydrocortisone

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups, whether using hydrocortisone or not during peri-operation, in parallel for the duration of the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, investigator, and outcome assessors are all prevented from having knowledge of the interventions assigned to individual participants. Care provider knows the individualized interventions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrocortisone withholding group (Experimental): Patients receive no hydrocortisone
  Interventions: Drug: Normal saline
- Hydrocortisone group (Active Comparator): Patients receive routine hydrocortisone
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Normal saline — No hydrocortisone or other steroids are given before, during, and after the surgery, except that patients develop postoperative adrenal insufficiency. If a patient develops postoperative adrenal insufficiency, he/she needs to receive hydrocortisone treatment (20mg at 0800 and 20mg at 1600) for one month and then check the level of morning serum cortisol to decide if it is time to start the hydrocortisone taper program.
  Other Names: Intravenous normal saline
  Arms: Hydrocortisone withholding group
Drug: Hydrocortisone — Hydrocortisone sodium succinate is given on the operation day (100mg at 0800 & 100mg at 2000), the postoperative day 1 (100mg at 0800 & 50mg at 2000), and the postoperative day 2 (25mg at 0800). Hydrocortisone (po.) is then given starting from the afternoon of postoperative day 2 (20mg at 1600 and 0800) to the end of the first postoperative week, and 20mg at 0800 during the second postoperative week. This is called the "hydrocortisone taper program". If a patient develops postoperative adrenal insufficiency, he/she needs to receive hydrocortisone treatment (20mg at 0800 and 20mg at 1600) for one month and then check the level of morning serum cortisol to decide if it is time to start the hydrocortisone taper program.
  Other Names: Hydrocortisone sodium succinate (iv.) & Hydrocortisone (po.)
  Arms: Hydrocortisone group

SUMMARY:
The investigators hypothesize that withholding hydrocortisone during the peri-operation in patients with pituitary adenomas whose hypothalamus pituitary adrenal axis are intact are safe.

DETAILED DESCRIPTION:
Pituitary is the headquarters of the endocrine system of the body, secreting several hormones maintaining the normal function of the endocrine organs. After surgery, pituitary dysfunction is seen in a small proportion of patients, even in some patients resulting in severe consequence, i.e. adrenal insufficiency or pituitary crisis. Therefore, patients undergoing pituitary surgery have been usually given "stress dose" steroids whether their hypothalamus pituitary adrenal (HPA) axis are deficient or preserved.

Results of several retrospective studies showed that there was no significantly increase in postoperative adrenal insufficiency in no supplementation (of hydrocortisone) group than in supplementation group. Given the considerable side effects of using steroids, whether hydrocortisone administration is necessary for all patients with pituitary adenomas during peri-operation needs to be discussed.

For Chinese patients with pituitary adenomas except for those of Cushing's disease, hydrocortisone administration during the peri-operation is a routine practice. Peking Union Medical College Hospital is the China Pituitary Disease Registry Center. Here, the investigators aim to launch a single-center prospective randomized controlled trial to verify the hypothesis that withholding hydrocortisone during the peri-operation in patients with pituitary adenomas whose HPA axis are intact are safe.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pituitary adenomas that need surgical resection of the tumor, whose hypothalamus-pituitary-adrenal axis are intact
* Patients of either gender aged from 18 years to 70 years

Exclusion Criteria:

* Patients with Cushing's disease
* Patients with pituitary adenomas who have already developed secondary adrenal insufficiency before surgery
* Patients with pituitary apoplexy or other acute pituitary conditions that need emergency surgery
* The postoperative pathology result indicates that the tumor is not a pituitary adenoma
* Patients that refuse to participate in the study or those who ask to quit after enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Rate of newly-onset adrenal insufficiency | During the first 3 postoperative days
  Adrenal insufficiency: lower-than-normal serum cortisol level at 8 a.m., plus the following related symptoms, including serious fatigue, muscle weakness, decreased appetite, nausea, vomiting, diarrhea, low blood pressure, palpitation, and fever.

SECONDARY OUTCOMES:
Rate of newly-onset adrenal insufficiency | From the 3rd postoperative day to the 3rd postoperative month
  Adrenal insufficiency: lower-than-normal serum cortisol level at 8 a.m., plus the following related symptoms, including serious fatigue, muscle weakness, decreased appetite, nausea, vomiting, diarrhea, low blood pressure, palpitation, and fever.

OTHER OUTCOMES:
Rate of newly-developed diabetes mellitus | During the first 3 postoperative months
  A random reading of blood sugar level more than 200 mg/dL (11.1 mmol/L), or a reading after two hours (after OGTT) over 200 mg/dL (11.1 mmol/L) indicates diabetes mellitus.
Rate of newly-developed diabetes insipidus | During the first 3 postoperative months
  Urine volume > 300ml for more than 3h or > 6 liter per day, specific gravity of urine <1.003, and serum sodium levels > 145 mmol/L indicate diabetes insipidus.
Concentration of blood electrolytes | At the 3rd postoperative month
  The level of Na+, K+, and Ca++ in the blood
Concentration of blood cells | At the 3rd postoperative month
  Numbers of erythrocytes, leukocytes, neutrophils, lymphocytes, thrombocytes in the blood
Percentage of blood cells | At the 3rd postoperative month
  Percentage of neutrophils, monocytes, lymphocytes of the leukocytes
Concentration of indexes of coagulation function #1 | At the 3rd postoperative month
  Prothrombin time, activated partial thromboplastin time, and thrombin time
Level of international normalized ratio | At the 3rd postoperative month
  Level of international normalized ratio
Level of D-Dimer | At the 3rd postoperative month
  Level of D-Dimer
Rate of deep venous thrombosis | During the first 3 postoperative months
  Deep venous thrombosis as detected by ultrasound
Rate of other complications | During the first 3 postoperative months
  Decreased bone density, osteoporosis, fracture, acne, and infections.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xing, MD, Study Chair — Neurosurgery, Peking Union Medical College Hospital, Beijing, China; Wei Lian, MD, Study Director — Neurosurgery, Peking Union Medical College Hospital, Beijing, China
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The individual participant data will be available upon reasonable requests to the study chair, Dr. Bing Xing, or the study director, Dr. Wei Lian.

REFERENCES:
- [Background] Tohti M, Li J, Zhou Y, Hu Y, Yu Z, Ma C. Is peri-operative steroid replacement therapy necessary for the pituitary adenomas treated with surgery? A systematic review and meta analysis. PLoS One. 2015 Mar 16;10(3):e0119621. doi: 10.1371/journal.pone.0119621. eCollection 2015. PMID 25775019
- [Background] Sterl K, Thompson B, Goss CW, Dacey RG, Rich KM, Zipfel GJ, Chicoine MR, Kim AH, Silverstein JM. Withholding Perioperative Steroids in Patients Undergoing Transsphenoidal Resection for Pituitary Disease: Randomized Prospective Clinical Trial to Assess Safety. Neurosurgery. 2019 Aug 1;85(2):E226-E232. doi: 10.1093/neuros/nyy479. PMID 30325449
- [Background] Lee HC, Yoon HK, Kim JH, Kim YH, Park HP. Comparison of intraoperative cortisol levels after preoperative hydrocortisone administration versus placebo in patients without adrenal insufficiency undergoing endoscopic transsphenoidal removal of nonfunctioning pituitary adenomas: a double-blind randomized trial. J Neurosurg. 2020 Jan 24;134(2):526-534. doi: 10.3171/2019.11.JNS192381. Print 2021 Feb 1. PMID 31978882
- [Derived] Guo X, Zhang D, Pang H, Wang Z, Gao L, Wang Y, Ma W, Lian W, Xing B; ZS-2608 Trial Team. Safety of Withholding Perioperative Hydrocortisone for Patients With Pituitary Adenomas With an Intact Hypothalamus-Pituitary-Adrenal Axis: A Randomized Clinical Trial. JAMA Netw Open. 2022 Nov 1;5(11):e2242221. doi: 10.1001/jamanetworkopen.2022.42221. PMID 36383383